CLINICAL TRIAL: NCT00416273
Title: Consolidation Therapy With Bortezomib <= 60 Year Old Patients With Multiple Myeloma
Brief Title: A Study of Bortezomib as Consolidation Therapy in Patients With Multiple Myeloma
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Janssen-Cilag G.m.b.H (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CR006124; 26866138MMY3012 (Other: Janssen-Cilag G.m.b.H, Germany); 2005-004948-31 (EudraCT Number)
Record Dates: First submitted 2006-12-22; First posted 2006-12-27 (Estimated); Last update posted 2015-03-06 (Estimated); Status verified 2015-03

CONDITIONS: Multiple Myeloma
Keywords: Multiple Myeloma; Bortezomib; PS341; Proteasome inhibitor; Consolidation therapy
MeSH Terms: conditions — Multiple Myeloma | interventions — Bortezomib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Treatment group (Experimental): Participants in the treatment group will receive Bortezomib at a dosage of 1.6 mg/m2.
  Interventions: Drug: Bortezomib
- Observation group (Experimental): Participants in the observation group will not receive any consolidation therapy.
  Interventions: Drug: No intervention

INTERVENTIONS:
Drug: Bortezomib — Bortezomib will be administered as 1.6 mg/m2 per body surface area on the days 1, 8, 15, 22 for the duration of 4 therapy cycles.
  Arms: Treatment group
Drug: No intervention — Participants in the observation group will be observed and will not receive any consolidation therapy.
  Arms: Observation group

SUMMARY:
The purpose of this study is determination of the event-free survival with and without Bortezomib consolidation therapy from the day of the first chemotherapeutic, myeloma-specific therapy measure, up to the occurrence of progression/recurrence or up to the occurrence of death.

DETAILED DESCRIPTION:
This is a two-arm (group), open-label (all people know the identity of the intervention), prospective (a study in which the patients are identified and then followed forward in time for the outcome of the study) randomized (the study medication is assigned by chance), multi-center study. Approximately 385 patients will be enrolled in this study. Patients will be randomly assigned to treatment or observation group in a ratio of 1:1. The study duration from screening up to the study end is up to 27 weeks. Then the patients will be observed until the last included patient has completed a 30 month post observational phase. The patients in the treatment arm will receive 4 cycles of a therapy. Each cycle lasts for a 35 days. Safety evaluations will include assessment of adverse events, vital signs, physical examination, electrocardiograms, and clinical laboratory tests.

ELIGIBILITY:
Inclusion Criteria:

* Patients with multiple myeloma with prior therapy consisting of remission induction therapy and high dose chemotherapy followed by stem cell transplantation
* Women must be postmenopausal or using safe contraception methods
* Creatinin clearance has to be higher than 30 ml/min and whole blood count has to be within acceptable ranges

Exclusion Criteria:

* No asecretory multiple myeloma
* History of allergic reactions to bortezomib or mannitol
* Expected life expectancy of less than 3 months
* No other malignant disease beside basalioma either existing or history of
* No history of severe cardio-pulmonary disease
* Seizures

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 217 (Actual)
Dates: Start 2006-12; Primary Completion 2013-05 (Actual); Study Completion 2013-05 (Actual)

PRIMARY OUTCOMES:
Number of patients with event-free survival (PFS) | From date of first chemotherapeutic myeloma-specific treatment measure until date of disease progression or death, whichever occurred first, as assessed approximately 30-60 months after the last patient was enrolled

SECONDARY OUTCOMES:
Number of patients with event free survival (EFS) | From date of first chemotherapeutic myeloma-specific treatment measure until the occurrence of the beginning of a new chemotherapeutic therapy,or death, whichever occurred first, as assessed approximately 30-60 months after the last patient was enrolled
Response rates | Up to Week 25
  Response will be determined according to EBMT (European Group for Blood and Marrow Transplantation) criteria; VGPR (very good partial response) will be added as an additional response criteria. VGPR is measured as at least 90 percents reduction of the monoclonal protein in the serum over at least 6 weeks.
Overall survival | From date of first chemotherapeutic myeloma-specific treatment measure until date of disease progression or death, whichever occurred first, as assessed approximately 30-60 months after the last participant was enrolled
  Time interval in months between the date of randomization and the participant's death from any cause.
Time to progression | From date of first chemotherapeutic myeloma-specific treatment measure until date of disease progression or death, whichever occurred first, as assessed approximately 30-60 months after the last participant was enrolled
  Time to progression is time interval in months until progression of disease, censoring for death or drop-out without progression.
Duration of response | Up to Week 25
  Duration of the response, measured from the day on which a response (at least minimal response) was documented for the first time after the start of the therapy, up until the day of the documentation of a progression/recurrence requiring therapy.
Number of patients with toxicities over the treatment period | Up to Week 24
  Toxicities will be assessed according to National Cancer Institute-Common Terminology Criteria for Adverse Events (NCI-CTCAE), version 3.
Change From Baseline in European Organization for Research and Treatment of Cancer quality of life questionnaire (EORTC QLQ-C30) | Baseline (Day 1), Enpoint (30-60 months)
  EORTC QLQ-C30 is a questionnaire to assess quality of life of cancer patients. It is composed of 30 items, multi-item measure (28 items) and 2 single-item measures. For the multiple item measure, 4-point scale is used and the score for each item range from "1 = not at all" to "4 = very much". Higher scores indicate worsening. The 2 single-item measure involves question about the overall health and overall quality of life which will be rated on a 7-point scale ranging from "1 = very poor" to "7 = excellent". Lower scores indicate worsening.
Number of the patients with skeletal related event (SRE) | Up to 30-60 months
  Pathological fracture, spinal cord compression, radiotherapy of a bone lesion, surgical therapy of a bone lesion will be considered as skeletal related events.
Time interval from the day of the transplantation up to the occurrence of the first SRE | Up to 30-60 months
Change From Baseline in EuroQol-5 (EQ-5D) Health Status Index to end point (30-60 months) | Baseline (Day 1) and end point (30-60 months)
  Change from Baseline to end point (30-60 months) in Euro Quality of life (Qol)-5 Dimension Questionnaire (EQ-5D). A higher score indicates an improvement in health in the Health Status Index. The EuroQol-5 is a five dimensional health state classification. Each dimension is assessed on a 3-point ordinal scale (1=no problems, 2=some problems, 3=extreme problems). The responses to the five EQ-5D dimensions were scored using a utility-weighted algorithm to derive an EQ-5D health status index score between 0 to 1, with 1.00 indicating "full health" and 0 representing dead.

CONTACTS AND LOCATIONS:
Overall Officials: Janssen-Cilag G.m.b.H, Germany Clinical Trial, Study Director — Janssen-Cilag G.m.b.H
Locations (38):
- Germany (38):
  - Augsburg
  - Bamberg
  - Berg
  - Berlin
  - Bremen
  - Cologne
  - Dresden
  - Duisburg
  - Erlangen
  - Eschweiler
  - Frankfurt am Main
  - Freiburg im Breisgau
  - Goch
  - Göttingen
  - Greifswald
  - Halle
  - Hamburg
  - Hamm
  - Hanover
  - Homburg
  - Jena
  - Karlsruhe
  - Kempten
  - Kiel
  - Magdeburg
  - Mainz
  - Mutlangen
  - München
  - Münster
  - Nuremberg
  - Oldenburg
  - Regensburg
  - Rostock
  - Stuttgart
  - Ulm
  - Villingen-Schwenningen
  - Wiesbaden
  - Würzburg

REFERENCES:
- [Derived] Straka C, Knop S, Vogel M, Muller J, Kropff M, Metzner B, Langer C, Sayer H, Jung W, Durk HA, Salwender H, Wandt H, Bassermann F, Gramatzki M, Rosler W, Wolf HH, Brugger W, Fischer T, Liebisch P, Engelhardt M, Einsele H. Bortezomib consolidation following autologous transplant in younger and older patients with newly diagnosed multiple myeloma in two phase III trials. Eur J Haematol. 2019 Sep;103(3):255-267. doi: 10.1111/ejh.13281. Epub 2019 Jul 19. PMID 31231828
- [Derived] Einsele H, Knop S, Vogel M, Muller J, Kropff M, Metzner B, Langer C, Sayer H, Jung W, Durk HA, Salwender H, Wandt H, Bassermann F, Gramatzki M, Rosler W, Wolf HH, Brugger W, Engelhardt M, Fischer T, Liebisch P, Straka C. Response-adapted consolidation with bortezomib after ASCT improves progression-free survival in newly diagnosed multiple myeloma. Leukemia. 2017 Jun;31(6):1463-1466. doi: 10.1038/leu.2017.83. Epub 2017 Mar 15. No abstract available. PMID 28293022
- See also: Consolidation Therapy with Bortezomib <= 60 Year Old Patients with Multiple Myeloma — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_JNJ_6051&studyid=242&filename=CR006124_CSR.pdf